CLINICAL TRIAL: NCT04364503
Title: Use of Patient Samples and Corresponding Clinical Data for Research and Development Studies And/or Population-based Analysis
Brief Title: Compliant Analysis of Patient Samples and Data
Status: Recruiting | Type: Observational
Sponsor: Sequenom, Inc. (Industry)
Collaborators: Laboratory Corporation of America (Industry)
Responsible Party: Sponsor
Other Study IDs: SCMM-RND-402
Record Dates: First submitted 2020-04-22; First posted 2020-04-28 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Pregnancy Related; Cancer; Infectious Disease
MeSH Terms: conditions — Neoplasms; Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Commercial remnant samples stored at multiple LabCorp affiliates.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Multiple interventions depending on diagnostic test being run. — Remnant samples and corresponding data from multiple diagnostic tests will be stored for future research and development.

SUMMARY:
Patients of scientific interest who have provided a commercial sample to LabCorp or one of its' affiliates will have their de-identified remnant samples and/or data used for research and development. Other commercial patients will be followed up on after informed consent is obtained.

DETAILED DESCRIPTION:
Arm 1 - Remnant commercial samples and data that has been de-identified of personal health information in compliance with HIPAA may be used for R&D studies or population-based analysis by LabCorp or affiliates.

Arm 2 - Collection of samples and/or data from commercial test patients requiring follow-up or from subjects of scientific interest after informed consent is obtained.

ELIGIBILITY:
Inclusion Criteria:

* Arm 1
* All samples and data are de-identified and HIPAA compliant
* Arm 2
* Subject is of scientific interest to the Sponsor or treating physician
* Subject provides written informed consent and has a clinical sample and/or supporting clinical data collected.

Exclusion Criteria:

* Arm 1
* Subject is from a US state or a country where local law restricts the use of de-identified data and/or remnants of specimens for research and/or development
* Arm 2
* Any medical or mental condition that would interfere with the subjects' ability to willingly give written informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Arm 1 - Female or male patient samples submitted to Sequenom or LabCorp affiliate for routine clinical care testing that no longer need to be maintained for clinical purposes.
  Arm 2 - Female or male subjects of scientific interest who have provided written informed consent/assent.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2018-03-17 (Actual); Primary Completion 2030-03-17 (Estimated); Study Completion 2030-08-15 (Estimated)

PRIMARY OUTCOMES:
Remnant samples and data for research and development | Retrospective and Prospective collection. Samples and data may be collected for up 12 months after enrollment.
  Remnant samples and data for research and development
Sample and data collection from subjects of scientific interest | Prospective collection. Samples and data may be collected for up to 12 months after enrollment
  Collect additional clinical data and samples if needed from subjects tested by LabCorp or an affiliate.

CONTACTS AND LOCATIONS:
Overall Officials: Graham P McLennan, Principal Investigator — Sequenom, Inc.
Locations (1):
- Sequenom, Inc, San Diego, California, United States